CLINICAL TRIAL: NCT05069974
Title: Oral and Neuro-Penetrative Alternative Antibiotics for Patients With Syphilis
Brief Title: Alternative Antibiotics for Syphilis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Principal Investigator, Oriol Mitja, Principal Investigator, Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trep-AB; 2020-005604-19 (EudraCT Number)
Record Dates: First submitted 2021-09-16; First posted 2021-10-06 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Early Latent Syphilis; Primary Syphilis; Secondary Syphilis
Keywords: Syphilis; Benzathine penicillin G; RPR; Treponema pallidum; Linezolid
MeSH Terms: conditions — Syphilis, Latent; Syphilis, primary; Syphilis, secondary; Syphilis; Treponemal Infections | interventions — Linezolid

STUDY DESIGN:
Intervention Model Description: Open-label, non inferiority, randomized clinical trial. Eligible patients will be randomized to recieve Linezolid (experimental arm) or BPG (control arm).
Who Masked: Outcomes Assessor
Masking Description: The statistical analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Linezolid (LZD) 1200 (Experimental): Patients will take film coated tables of LZD 600 mg every 12 hours during 10 days
  Interventions: Drug: Linezolid 600 mg
- Benzathine Penicillin G (BPG) (Active Comparator): Administration of intramuscular BPG 2.4 MIU single dose during day 1
  Interventions: Drug: Benzathine Penicilllin G
- Linezolid (LZD) 600 (Experimental): Patients will take film coated tables of LZD 600 mg every 24 hours during 5 days
  Interventions: Drug: Linezolid 600 mg

INTERVENTIONS:
Drug: Linezolid 600 mg — After randomized to the experimental arm, the patient will take 1 tablet of Linezolid every 12hours during 10 days or 1 tablet of of Linezolid every 24hours during 5 days.
  Arms: Linezolid (LZD) 1200; Linezolid (LZD) 600
Drug: Benzathine Penicilllin G — After randomized to the control arm, the patient will receive a single dose of intramuscular BPG.
  Arms: Benzathine Penicillin G (BPG)

SUMMARY:
The Trep-AB clinical trial will test the efficacy of an investigational neuropenetrative drug, Linezolid (LZD), compared to standard treatment, Benzathine penicillin G (BPG), for early syphilis in humans. The overarching idea of the work proposed herein is to investigate the use of LZD to treat syphilis, conducting a randomized controlled clinical trial to evaluate this new indication of a known antibacterial agent.

DETAILED DESCRIPTION:
The syphilis epidemic is rampant around the world, and therapeutic options are restricted to an antibiotic, intramuscular (IM) BPG, which does not efficiently cross the blood-brain barrier. Treponema pallidum (T.p.), the bacteria that causes syphilis, invades the central nervous system (CNS) in 40% of patients, usually without symptoms. The prognostic implications of CNS invasion are the potential for severe neurologic complications, and treatment failure due to sequestered bacteria in the CNS. When indicated, the only way to identify and treat neurosyphilis is by lumbar puncture to examine the cerebrospinal fluid (CSF), followed by intravenous (IV) Benzyl penicillin therapy. The invetigators have carried out in silico studies showing that oxazolidinones are potentially active against T.p., are neuropenetrative and can be administered orally. The invetigators have carried out preclinical studies using an in vitro culture system for T.p. and the use of the syphilis animal model with rabbits to test different antibiotics. The invetigators have confirmed that LZD was the best compound that could go on to be tested in clinical trials to treat syphilis.

The Trep-AB clinical trial will test the efficacy of an investigational neuropenetrative drug, LZD, compared to standard treatment BPG, for early syphilis in humans conducting a randomized controlled clinical. Primary objective is to demonstrate the non-inferiority of LZD treatment compared with standard BPG treatment to cure patients with early syphilis. Seconday objective is to isolate T.p. strains in clinical samples to subtype DNA from patients at baseline and during recurrence or treatment failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at baseline visit.
2. Primary, secondary or early latent syphilis diagnosis based on SEIMC/IUSTI Guidelines*

   1. Primary syphilis is defined as typical ulcer (chancre) and positive test using darkfield examination (DFE) or Polymerase chain reaction (PCR) detection of T.p. with/without positive serological test for syphilis.
   2. Secondary syphilis is defined based on typical clinical symptoms with positive treponemal and non-treponemal tests.
   3. Early latent syphilis is defined as positive serological treponemal and non-treponemal tests with no clinical evidence of infection, with a previous negative syphilis serology,or a four-fold increase in RPR titer of a non-treponemal test within the past 12 months.Serological tests for syphilis performed within 10 days prior to study inclusion visit willbe acceptable for enrollment.
3. Signature of written informed consent.
4. Ability to comply with the requirements of the study protocol.
5. If women of childbearing potential, use of a highly effective method of contraception (abstinence,hormonal contraception, intra-uterine device [IUD], or anatomical sterility in self or partner)committed during 1 week after last IMP administration.
6. If men, use of condom during heterosexual intercourse and use of a highly effective method ofcontraception (abstinence, hormonal contraception, intra-uterine device [IUD], or anatomical sterilityin self or partner) in female partner committed during 1 week after last IMP administration.

   * For inclusion purposes, positive point of care tests (POCT) will be accepted in selected patients without previous syphilis history and negative serological tests for syphilis during the last 12 months (Syphilis rapid diagnostic test [RDT] or Chembio DPP syphilis screen & confirm assay [DPP]), or with a previous history of syphilis and negative non-treponemal tests during the last 12 months (DPP). Further confirmation by the methods described in a), b) or c) will benecessary.

Exclusion Criteria:

1. Known allergy to any of the IMPs and/or excipients, particularly known hypersensitivity to penicillin, cephalosporins or other beta-lactam agents and/or allergy to soya or peanut.
2. Lactose or galactose intolerance or glucose-galactose malabsorbtion.
3. Diagnosis criteria of symptomatic neurosyphilis.
4. Pregnant or breastfeeding women.
5. Current treatment with any drugs likely to interact with the study medication (see Appendix 6).
6. Have taken any antibiotics with potential activity against syphilis (e.g. beta lactams, cephalosporines, macrolides, tetracyclines) within 1 week prior to randomization.
7. Uncontrolled hypertension, pheochromocytoma, thyrotoxicosis, carcinoid syndrome, bipolar disorder, incapacitating psycho-affective disturbance, acute confusional state.
8. Renal function impairment requiring hemodialysis.
9. Symptomatic concomitant STI (i.e., gonococcus, chlamydia, lymphogranuloma venereum, Mycoplasma genitalium) or other infection disease requiring antibiotic treatment potentially active against syphilis.
10. Having received treatment for the early syphilis recently diagnosed (In the previous 6 months)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with clinical resolution of primary syphilis lesions (clinical cure, primary). | at week 2
  Assesment of clinical resolution defined as the complete healing of primary syphilis lesions within 2 weeks from treatment start.
Proportion of patients with clinical resolution of secondary syphilis lesions (clinical cure, secondary). | at week 6
  Assesment of clinical resolution defined as the complete healing of secondary syphilis lesions within 6 weeks from treatment start.
Proportion of patients with adequate serological response (serological cure, week 12). | at week 12
  Assessment of adequate serological response defined as a four-fold decline in rapid plasma reagin (RPR) titer or seroreversion to negative.
Proportion of patients with adequate serological response (serological cure, week 24). | at week 24
  Assessment of adequatesserological response defined as a four-fold decline in rapid plasma reagin (RPR) titer or seroreversion to negative.
Proportion of patients with adequate serological response (serological cure, week 48). | at week 48
  Assessment of adequate serological response defined as a four-fold decline in rapid plasma reagin (RPR) titer or seroreversion to negative.
Proportion of patients with allelic variation in T. pallidum strain(s) DNA in recurrent syphilis or suspected treatment failure (molecular cure). | From date of randomization until date of first documented recurrence or treatment failure, assesed up to 48 weeks
  Assessment of re-infection in recurrent syphilis as defined by allelic variation in core genes of T. pallidum strain(s) compared to baseline using a molecular method (MLST-WGS).

SECONDARY OUTCOMES:
Proportion of patients with allelic variation in T. pallidum strain(s) DNA in ulcer or mucosa lesions swabs (re-infection). | From date of randomization until date of first documented recurrence, assesed up to 48 weeks
  Assessment of re-infection in recurrent syphilis lesions as defined by allelic variation in core genes of T. pallidum strain(s) compared to baseline using a molecular method (MLST-WGS).
Proportion of patients with allelic variation in T. pallidum strain(s) DNA in plasma (re-infection). | From date of randomization until date of first documented recurrence, assesed up to 48 weeks
  Assessment of re-infection in recurrent syphilis (secondary or early latent) as defined by allelic variation in core genes of T. pallidum strain(s) compared to baseline using a molecular method (MLST-WGS).
Proportion of patients with allelic variation in T. pallidum strain(s) DNA in oral swab/saliva (re-infection). | From date of randomization until date of first documented recurrence, assesed up to 48 weeks
  Assessment of re-infection in recurrent syphilis (secondary or early latent) as defined by allelic variation in core genes of T. pallidum strain(s) compared to baseline using a molecular method (MLST-WGS).
Proportion of patients with allelic variation in T. pallidum strain(s) DNA in skin punch biopsy (re-infection). | From date of randomization until date of first documented recurrence, assesed up to 48 weeks
  Assessment of re-infection in recurrent syphilis lesions as defined by allelic variation in core genes of T. pallidum strain(s) compared to baseline using a molecular method (MLST-WGS).
Proportion of patients with allelic variation in T. pallidum strain(s) DNA in ear lobe scraping (re-infection). | From date of randomization until date of first documented recurrence, assesed up to 48 weeks
  Assessment of re-infection in recurrent syphilis (secondary or early latent) as defined by allelic variation in core genes of T. pallidum strain(s) compared to baseline using a molecular method (MLST-WGS). (Optional,in a selected group of patients).
Proportion of patients with suspicion of neurosyphilis that have allelic variation in Treponema pallidum (T.p) isolates DNA in CSF (re-infection). | From date of randomization until date of first documented recurrence, assesed up to 48 weeks
  Assessment of re-infection in patients with suspicion of neurosyphilis as defined by allelic variation in core genes of T. pallidum strains compared to baseline using a molecular method (MLST-WGS). (in a selected group of patients with suspicion of neurosyphilis).
Proportion of patients with antibiotic resistance genotype. | From date of randomization until date of first documented recurrence, assesed up to 48 weeks
  Assesment of allelic variation in core genes conferring antimicrobial resistance in clinical specimens from patients who are considered to have treatment failure compared to patients with adequate clinical and serological response.
Proportion of participants experiencing adverse events. | up to 12 weeks
  Assesment of adverse events related to LZD treatment compared with adverse events related to standard BPG treatment in participants with early syphilis.
Proportion of patients who have a change in the RPR titer within 2 weeks after treatment start of primary syphilis. | at 2 weeks
  Assessment of RPR titer variation at week 2 from treatment start of patients with primary syphilis.

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Mitjà Villar, PhD, Principal Investigator — Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Locations (6):
- Spain (5):
  - CAP Drassanes-Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Barcelona Checkpoint, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Germans Trias Pujol, Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid, Madrid
- Mortimer Market Centre, London, United Kingdom

REFERENCES:
- [Derived] Ubals M, Nadal-Baron P, Arando M, Rivero A, Mendoza A, Descalzo Jorro V, Ouchi D, Perez-Mana C, Alvarez M, Alemany A, Hoyos-Mallecot Y, Nunley E, Lieberman NAP, Greninger AL, Galvan-Casas C, Suner C, G-Beiras C, Paredes R, Rodriguez-Gascon A, Canut A, Garcia-Patos V, Farre M, Marks M, Giacani L, Vall-Mayans M, Mitja O. Oral linezolid compared with benzathine penicillin G for treatment of early syphilis in adults (Trep-AB Study) in Spain: a prospective, open-label, non-inferiority, randomised controlled trial. Lancet Infect Dis. 2024 Apr;24(4):404-416. doi: 10.1016/S1473-3099(23)00683-7. Epub 2024 Jan 8. PMID 38211601